CLINICAL TRIAL: NCT05003531
Title: A Phase II Multicenter, Randomized, Double-blind, Parallel, Placebo-controlled Trial to Evaluate the Efficacy and Safety of IBI112 in Different Dose Regimens for the Treatment of Subjects With Moderate-to-severe Plaque Psoriasis
Brief Title: A Study to Evaluate IBI112 in the Treatment of Subjects With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI112A201
Record Dates: First submitted 2021-08-05; First posted 2021-08-12 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- IBI112 dose 1 (Experimental): Participants will receive IBI112 dose 1 subcutaneous injection(SC)
  Interventions: Drug: IBI112 dose 1
- IBI112 dose 4 (Experimental): Participants will receive IBI112 dose 4 subcutaneous injection(SC)
  Interventions: Drug: IBI112 dose 4
- IBI112 dose 2 (Experimental): Participants will receive IBI112 dose 2 subcutaneous injection(SC)
  Interventions: Drug: IBI112 dose 2
- IBI112 dose 3 (Experimental): Participants will receive IBI112 dose 3 subcutaneous injection(SC)
  Interventions: Drug: IBI112 dose 3
- Placebo (Placebo Comparator): Participants will receive placebo subcutaneous injection(SC)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: IBI112 dose 2 — Participants will receive placebo or dose 2 IBI112 SC
  Arms: IBI112 dose 2
Drug: IBI112 dose 4 — Participants will receive placebo or dose 4 IBI112 SC
  Arms: IBI112 dose 4
Drug: IBI112 dose 1 — Participants will receive placebo or dose 1 IBI112 SC
  Arms: IBI112 dose 1
Drug: IBI112 dose 3 — Participants will receive placebo or dose 3 IBI112 SC
  Arms: IBI112 dose 3
Drug: placebo — Participants will receive placebo SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of IBI112 administered in different dose regimens for the treatment of patients with plaque psoriasis

ELIGIBILITY:
Inclusion criteria

* Diagnosis of plaque-type psoriasis with or without psoriatic arthritis for at least 6 months prior to first administration of any study agent
* Must be a candidate for phototherapy or systemic treatment for psoriasis (either new to treatment or having had previous treatment)

Exclusion criteria

* History of or current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease
* Participant has history of erythrodermic psoriasis, generalized or localized pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new onset guttate psoriasis
* Has received any therapeutic agent directly targeted to IL-12, IL-17, or IL-23within 6 months of the first administration of study agent
* Has received any therapeutic agent directly targeted toTNF-a within 3 months of the first administration of study agent
* Has received any conventional therapeutic agent within 1 months of the first administration of study agent
* Has received any topic therapeutic agent within 2 weeks of the first administration of study agent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving Psoriasis Area and severity index(PASI) 90 at week 16 | Week 16
  PASI 90 is defined as at least a 90% reduction in PASI relative to baseline

SECONDARY OUTCOMES:
Percentage of patients achieving Psoriasis Area and severity index(PASI) 75 at week 16 | Week 16
  PASI 75 is defined as at least a 75% reduction in PASI relative to baseline
Percentage of patients achieving Psoriasis Area and severity index(PASI) 100 at week 16 | Week 16
  PASI 100 is defined as at least a 100% reduction in PASI relative to baseline
Percentage of patients with Physician Global Assessment(PGA) Score of Cleared(0) or Minimal(1) at week 16 | Week 16
  PGA of psoriasis is used to determine the participant's psoriasis lesions overall at a given time point.PGA score ranges from 0-4,0=cleared, 1= minimal ,2=mild, 3= moderate, 4= marked, 5= severe
Percentage of patients with Physician Global Assessment(PGA) Score of Cleared(0) at week 16 | Week 16
  PGA of psoriasis is used to determine the participant's psoriasis lesions overall at a given time point.PGA score ranges from 0-4,0=cleared, 1= minimal ,2=mild, 3= moderate, 4= marked, 5= severe
Change from Baseline in Dermatology life quality index(DLQI) at week 16 | Week 16
  The DLQI is a 10-item questionnaire that measures the impact of skin disease on participant's quality of life
Percentage of patients achieving Psoriasis Area and severity index(PASI) 90 at week 52 | Week 52
  PASI 90 is defined as at least a 90% reduction in PASI relative to baseline
Percentage of patients achieving Psoriasis Area and severity index(PASI) 100 at week 52 | Week 52
  PASI 100 is defined as at least a 100% reduction in PASI relative to baseline
Percentage of patients achieving Psoriasis Area and severity index(PASI) 75 at week 52 | Week 52
  PASI 75 is defined as at least a 75% reduction in PASI relative to baseline
Percentage of patients with Physician Global Assessment(PGA) Score of Cleared(0) or Minimal(1) at week 52 | Week 52
  PGA of psoriasis is used to determine the participant's psoriasis lesions overall at a given time point.PGA score ranges from 0-4,0=cleared, 1= minimal ,2=mild, 3= moderate, 4= marked, 5= severe
Percentage of patients with Physician Global Assessment(PGA) Score of Cleared(0) at week 52 | Week 52
  PGA of psoriasis is used to determine the participant's psoriasis lesions overall at a given time point.PGA score ranges from 0-4,0=cleared, 1= minimal ,2=mild, 3= moderate, 4= marked, 5= severe
Change from Baseline in Dermatology life quality index(DLQI) at week 52 | Week 52
  The DLQI is a 10-item questionnaire that measures the impact of skin disease on participant's quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- PeKing University People's Hostpital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No